CLINICAL TRIAL: NCT07094386
Title: Ultrasound Guided Techniques for Postoperative Analgesia in Patients Undergoing Open Upper Abdominal Surgeries: External Oblique Intercostal Plane Block vs. Quadratus Lumborum Block; A Randomized Controlled Trial
Brief Title: Postoperative Analgesia in Patients Undergoing Open Upper Abdominal Surgeries: External Oblique Intercostal Plane Block vs. Quadratus Lumborum Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Shaaban Glall Ismail, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-135-2025
Record Dates: First submitted 2025-07-16; First posted 2025-07-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group External Oblique Intercostal Plain Block (EOIPB) (Active Comparator): Patients will receive general anesthesia initially then unilateral EOIPB with total volume 30 ml of bupivacaine 0.25% will be performed.
  Interventions: Procedure: External Oblique Intercostal Plain Block; Drug: Bupivacaine %0.25 (isobaric)
- Group Quadratus Lumborum Block (QLB) (Active Comparator): Patients will receive general anesthesia initially then unilateral QLB with total volume 30 ml of bupivacaine 0.25% will be performed.
  Interventions: Procedure: Quadratus Lumborum Block; Drug: Bupivacaine %0.25 (isobaric)

INTERVENTIONS:
Procedure: External Oblique Intercostal Plain Block — The patient will be placed in the supine position. After sterilization of the skin, a high-frequency linear probe (6-13 MHz) will be placed obliquely medial to the anterior axillary line, the 6th and 7th ribs, skin, subcutaneous tissues, and external oblique muscle [EOM], intercostal muscles, pleura, and the lung will be identified. An 80 mm 22-gauge block needle (Stimuplex® D, BBraun, Germany) will be inserted in-plane to the US-probe in a craniocaudal direction directed under EOM. After confirmation of negative blood aspiration, 2-3 mL of normal saline will be injected for hydro-dissection to verify the correct needle tip placement then 30 mL of 0.25% bupivacaine will be injected between the EOM and intercostal muscles
  Arms: Group External Oblique Intercostal Plain Block (EOIPB)
Procedure: Quadratus Lumborum Block — Quadratus lumborum block will be performed. The patient will be placed in the lateral decubitus position After sterilization of the skin, a low frequency convex probe (5-8 MHz) will be positioned horizontally in the anterior axillary line half way between the subcostal margin and the iliac crest then will be advanced in the cranial direction to visualize the triple abdominal muscle layers and identifying the posterior border of the EO muscle (hook sign) with the underlying IO musclenforming a roof over the QL muscle. The QL muscle could be visualized with its attachment to the lateral edge of the transverse process of the L4 vertebral body. An 80 mm 22-gauge block needle will be inserted in-plane to the US-probe in an anterolateral to posteromedial direction. The needle tip will be placed between the middle layer of the thoracolumbar fascia and the QL muscle. After confirmation of negative blood aspiration, 30 mL of 0.25% bupivacaine will be injected.
  Arms: Group Quadratus Lumborum Block (QLB)
Drug: Bupivacaine %0.25 (isobaric) — A single injection of 30 mg of 0.25 % bupivacaine will be administered as part of the External Oblique Intercostal Plain Block under ultrasound guidance, after confirming needle placement between the external oblique and intercostal muscles.
  Arms: Group External Oblique Intercostal Plain Block (EOIPB)
Drug: Bupivacaine %0.25 (isobaric) — A single injection of 30 mg of 0.25 % bupivacaine will be administered as part of the Quadratus Lumborum Block under ultrasound guidance, after confirming of correct needle placement and negative aspiration.
  Arms: Group Quadratus Lumborum Block (QLB)

SUMMARY:
Open upper abdominal surgeries with subcostal incisions are a cause of severe pain and can lead to pulmonary and cardiac complications, detrimental physiological effects, and may also have psychological, economic, and social adverse effects if inadequately treated. Effective pain control can avoid these complications and contribute to several clinically valuable outcomes, including earlier patient mobilization and quicker recovery, which can result in a shortened hospital stay and reduced costs.

Opioids are the gold standard in postoperative pain control. however, it increases the incidence of opioid related adverse events such as respiratory depression, dizziness, nausea, vomiting and constipation. Regional analgesia plays an important role in perioperative multimodal analgesic regimens for major abdominal surgeries. The ultrasound-guided technique provides several options for relieving postoperative pain.

The aim of this study is to compare the efficacy and safety of ultrasound guided external oblique intercostal plane block versus quadratus lumborum in patients undergoing open upper abdominal surgeries.

DETAILED DESCRIPTION:
Poorly controlled postoperative pain causes physiological stress, increased morbidity, delayed mobilization, prolonged hospitalization, and higher healthcare costs.

Regional anelgesia techniques have shown a promise in improving postoperative outcomes by reducing opioid consumption and related adverse effects.

This study aims to evaluate two regional blocks - EOIPB and QLB- both will be performed under ultrasound guidance.

The goal is to determine which technique offers superior analgesic efficacy, safety and overall contribution to the quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both sexes.
* 18 to 60 years old.
* ASA physical status I- III scheduled for elective open upper abdominal surgeries, as (open nephrectomy, open cholecystectomy, liver resection, ….).
* Patients with BMI (18.5-35) kg/ m2.

Exclusion Criteria:

* Patients uncooperative or refuse to sign the consent of regional block.
* Patients with known coagulation defects. International normalized ratio (INR)> 1.5), and thrombocytopenia if platelet count < 100.000).
* Patients with known hypersensitivity to bupivacaine, or any of the used drugs.
* Patients with hepatic impairment, as Child-Pugh class B or C, AST/ALT > 3 times the upper limit of normal, or total bilirubin > 2 mg/dL.
* Patients with renal impairment, chronic kidney disease stage 4 or 5 (eGFR < 30 mL/min/1.73 m²), or on regular dialysis.
* Patients with pre-existing myopathy, defined as a clinically diagnosed muscular disorder characterized by muscle weakness, elevated creatine kinase levels, or a history of inherited or acquired muscle disease (e.g., polymyositis, muscular dystrophy).
* Patients with pre-existing neuropathy, if clinically diagnosed as peripheral or central nerve dysfunction, including chronic sensorimotor deficits or conditions such as diabetic neuropathy, radiculopathy, or multiple sclerosis.
* Patients with chronic pain syndromes, defined as pain persisting for more than 3 months, including fibromyalgia, complex regional pain syndrome (CRPS), or chronic pain requiring long-term opioid or neuropathic pain medications.
* Patients with sepsis at the site of injection.
* Patients with history of long-acting opioids or steroids preoperatively

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Time to first requested rescue analgesia (minutes) | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Nesrine Elrefai, Professor, Study Director — Cairo university, Faulty of Mdicine; Ahmed El Sakka, Professor, Study Chair — Cairo university, Faulty of Mdicine
Locations (1):
- Cairo university hospitals, Cairo, Egypt